CLINICAL TRIAL: NCT03990142
Title: Study of Abnormalities of the Vegetative Nervous System in the Occurrence of Intradialytic Arterial Hypotension
Brief Title: Study of Abnormalities of the Nervous System in the Occurrence of Intradialytic Arterial Hypotension
Acronym: SUDHEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUDHEMO
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Intervention Model Description: Patients will be classified into 2 groups according to the occurrence of intradialytic hypotension which is defined as a decrease in systolic blood pressure greater than 30 mmHg associated with clinical signs (cramps, abdominal pain, unconsciousness, convulsions). Group 1 corresponds to patients with intradialytic hypotension and group 2 corresponds to patients without intradialytic hypotension. This study aims to measure the cutaneous conductance to chlorine by SUDOSCAN® in all dialysis patients and to seek a link between the results of this examination and the occurrence of discomfort during hemodialysis sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: patients without intradialytic hypotension (Experimental): The investigators will measure the cutaneous conductance to chlorine by SUDOSCAN® in all dialysis patients without intradialytic hypotension and to seek a link between the results of this examination and the occurrence of discomfort during hemodialysis sessions.
  Interventions: Diagnostic Test: Cutaneous conductance to chlorine by SUDOSCAN
- Group 2: patients with intradialytic hypotension (Experimental): The investigators will measure the cutaneous conductance to chlorine by SUDOSCAN® in all dialysis patients with intradialytic hypotension and to seek a link between the results of this examination and the occurrence of discomfort during hemodialysis sessions.
  Interventions: Diagnostic Test: Cutaneous conductance to chlorine by SUDOSCAN

INTERVENTIONS:
Diagnostic Test: Cutaneous conductance to chlorine by SUDOSCAN — The additional examination, related to this research protocol, corresponds to a record of cutaneous conductance with chlorine. This recording of 2 min 30 is done thanks to SUDOSCAN® within 30 minutes before the dialysis session (before the "connection" to the dialysis machine) and within 30 minutes after the end of the dialysis with a measurement of the tension blood pressure and heart rate immediately before SUDOSCAN®.

SUMMARY:
Intradialytic hypotension is a common complication of hemodialysis sessions in patients with chronic renal failure, with an estimated prevalence of 10 to 30%. This hypotensopn is classically defined by a decrease in systolic blood pressure greater than 30 mmHg associated with clinical signs (cramps, abdominal pain, unconsciousness, convulsions). Its repetition is correlated with cardiovascular events, neurological events and excess mortality. Several clinical factors have been proposed to predict the risk of intradialytic hypotension such as age, certain comorbidities (diabetes, ischemic heart disease...), dialysis modalities (hemodialysis), ultrafiltration, conductivity but also alterations of the autonomic nervous system (especially the sympathetic system).

In recent years, the study of vegetative functions has been facilitated by the use of SUDOSCAN® (Impeto, Paris, France) which is a simple, non-invasive tool that allows the study of Chlorine conductance directly reflecting the activity of small non-myelinated C fibers that innervate the sweat glands. SUDOSCAN® has shown good sensitivity and specificity in the diagnosis of vegetative damage in diabetic patients and also a good correlation with cardiac autonomic neuropathy. More recently, SUDOSCAN® has shown good sensitivity in the detection of neuropathies small fibers especially in diabetic patients. This sensitivity is comparable to QST-type quantitative tests and the correlation with cardiovascular dysautonomia tests is good. This test, simple and fast realization, does not require the active participation of the patient. There is a good correlation between the results of SUDOSCAN® and the reduction of intra-dermal fiber density at cutaneous biopsy.

Hemodialysis patients are at risk of peripheral neurological involvement not only because of an increasing incidence of diabetes (30-40%) but also because of the abnormal production and elimination of certain uremic toxins. Few studies exist on the anomalies of the vegetative system in hemodialysis. A recent publication has suggested a difference in nerve excitability depending on the type of hemodialysis suggesting nerve changes secondary to ionic changes. The identification of patients at risk of intradialytic hypotension during dialysis sessions could be useful for adapting hemodialysis protocols.

Patients will be classified into 2 groups according to the occurrence of intradialytic hypotension. Group 1 corresponds to patients with intradialytic hypotension and group 2 corresponds to patients without intradialytic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient on hemodialysis for more than 6 months
* Patient affiliated with a health insurance plan
* Francophone patient
* Patient giving free, informed and express consent

Exclusion Criteria:

* Patient with lesions, wounds, amputations preventing the measurement of the chlorine conductance of the palms of the hands and feet
* Patient with a disability that prevents them from standing while measuring conductance / SUDOSCAN®
* Patient already included in an interventional research protocol
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Cutaneous conductance to chlorine by SUDOSCAN before hemiodialysis | Day 1
  This outcome is to measure cutaneous conductance to chlorine by SUDOSCAN, 30 minuts before hemodialysis.

SECONDARY OUTCOMES:
Cutaneous conductance to chlorine by SUDOSCAN after hemiodialysis | Day 1
  This outcome is to measure cutaneous conductance to chlorine by SUDOSCAN, 30 minuts after hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline REACH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- AURA Paris Plaisance, Paris, France

REFERENCES:
- [Result] Reach P, Touzot M, Lombardi Y, Maheas C, Sacco E, Fels A, Beaussier H, Urena-Torres P, Chatellier G, Ridel C, Zuber M. Electrochemical skin conductance by Sudoscan(R): a new tool to predict intradialytic hypotension. Nephrol Dial Transplant. 2021 Jul 23;36(8):1511-1518. doi: 10.1093/ndt/gfab183. PMID 34021358